CLINICAL TRIAL: NCT02908555
Title: Sleep, Coping, and Executive Functioning in Youth With Type 1 Diabetes
Brief Title: Sleep, Coping and Executive Functioning in Youth With Type 1 Diabetes
Acronym: SleepT1D
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1507016174
Record Dates: First submitted 2016-09-08; First posted 2016-09-21 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; adolescents; sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no intervention: Descriptive study without groups
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a descriptive study with no intervention

SUMMARY:
The purpose of this exploratory study is to evaluate the characteristics of sleep, perceptions of barriers and facilitators to adequate sleep, and the associations among sleep characteristics, executive functioning, coping, adherence, 24-hour glucose levels, and adjustment in adolescents with type 1 diabetes. A mixed methods approach that includes a quantitative component, consisting of actigraphy and sleep diaries, questionnaires, tests of executive function and continuous glucose monitoring (CGM) as well as a narrative qualitative component will be used. Results from this pilot study will be used to provide the effect sizes needed for a larger-scale descriptive study and to establish the need for a possible sleep-promoting intervention for adolescents with type 1 diabetes. This project is consistent with ongoing research focused on developing preventive, behavioral interventions for youth with type 1 diabetes and their families to improve physiological (i.e., glycemic control) and psychological (i.e., quality of life) outcomes. Sleep promotion may become an important component of these interventions. Thus, the following specific aims will be addressed:

1. Describe the objective and subjective characteristics of sleep (duration, continuity, bed time/rise times); sleep quality and sleep habits among adolescents with type 1 diabetes.
2. Explore the relationship between characteristics of self-reported sleep (i.e., habits, duration, daytime sleepiness) and executive function, coping, adherence, and adjustment (i.e., depressive symptoms, quality of life) in adolescents with type 1 diabetes.
3. Explore the relationship of glucose excursions on sleep characteristics and executive functioning.

3. Conduct a qualitative study using narrative analysis with adolescents to identify perceived barriers, facilitators, and consequences associated with insufficient sleep in adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
A mixed methods approach will be used to characterize sleep and explore the associations between sleep disturbances and executive function, coping, glycemic control, adherence, and adjustment in adolescents with type 1 diabetes. To understand these relationships, the investigators will collect quantitative data, including self-report and parent-report questionnaires and a test of cognitive functioning after consent and screening. Clinical data related to diabetes will be collected from the medical chart and CGM, and overnight sleep data will be collected during the subsequent week. The investigators will also collect qualitative data, using semi-structured interviews.

Aim 1. Describe the objective and subjective characteristics of sleep (duration, continuity, bed time/rise times); sleep quality and sleep habits among adolescents with type 1 diabetes.

After completing the initial recruitment procedures and questionnaires, adolescents will wear the Respironics Minimitter Actiwatch AW64, a wrist-worn accelerometer, continuously for 1 week, removing them only for bathing, and depress the event marker at "lights out" and "lights on" times to demarcate time in bed. Sleep diaries will be completed daily in the mornings and evenings to track daytime sleep-related behaviors (e.g., caffeine use, exercise) and nocturnal sleep characteristics (e.g., bedtime, wakings). The research assistants will call adolescents the day after enrollment to address any problems and elicit understanding. At the end of the week, they will call adolescents as a reminder to complete the data collection and return the watch and diary in a prepaid mailer.

Data Analysis. Actigraph data will be scored with Actiware v. 5 software. Diary forms have been prepared in scannable format to reduce the need for research staff entering data manually. Forms will be examined for improperly filled items and missing data, scanned and committed to an MS Access database. Descriptive statistics will be used to summarize each of the primary sleep variables (diary and actigraph) (% wake after sleep onset, time in bed, sleep efficiency, sleep latency, duration) over the 1-week interval. Descriptive statistics will also be used to characterize the total and component scores of the Children's Sleep Questionnaire.

The expected outcome of this aim is a more detailed characterization of sleep patterns in adolescents with T1D to identify the key variables to be measured in a large scale study.

Aim 2. Explore the relationship between characteristics of self-reported sleep (i.e., habits, duration, daytime sleepiness) and executive function, coping, adherence, and adjustment (i.e., depressive symptoms, quality of life, anxiety) in adolescents with type 1 diabetes. Questionnaires and test of executive function will be completed by adolescents and their parent/guardian after screening and consent.

Measures: The proposed measures have been used in our ongoing studies with adolescents with T1D, and they have established reliability and validity. The questionnaires will take about 20-30 minutes to complete, and the test of executive function will take 5 minutes. Following the established protocol, a trained RA will demonstrate the Trail Making Test using the sample sheet. The adolescent will be timed on the full test (drawing lines to connect 25 circles, alternating letters and numbers).

Data Analysis: To explore the relationship between sleep and executive function, coping, adherence, and adjustment, the investigators will use bivariate correlations. To evaluate the extent to which insufficient sleep is associated with executive function, coping, adherence, and adjustment in this population the investigators will use conduct independent groups t-tests to obtain estimates of the differences on key variables between adolescents who get insufficient vs. sufficient sleep (< 7 hours/night vs. > 7 hours/night). The investigators will also calculate the effect size from these data to establish the basis for a power analysis for a possible future larger study. Finally, using a linear regression model, the effect of sleep duration on key variables will be examined after controlling for potential confounders; gender, race/ethnicity, and income have been shown to impact sleep habits. Further, the investigators will explore the extent to which there is an effect of gender on the outcome variables or their interactions.

The expected outcome of this aim is estimates of effect sizes needed to conduct power analyses for a full-scale study of the associations between sleep and cognitive function, coping, adherence, and adjustment.

Aim 3. Explore the relationship of glucose excursions on sleep characteristics and executive function. Using CGM data from the iPro CGM system, glucose excursions and time with hypoglycemia or hyperglycemia will be identified. Youth who are already using CGM will not have to wear a second monitor, but will provide downloaded data from their CGM at the return visit.

Data analyses: Bivariate correlations to examine relationships among sleep and executive function, coping, adherence, and adjustment and glycemic excursions will be conducted. To evaluate the extent to which insufficient sleep is associated with executive function, coping, adherence, and adjustment in this population independent groups t-tests will be used to obtain estimates of the differences on key variables between adolescents with nighttime hypo- or hyperglycemia. The effect size will be calculated from these data to establish the basis for a power analysis for a possible future larger study. Finally, using a linear regression model, the effect of sleep duration on key variables will be examined after controlling for potential confounders; gender, race/ethnicity, and income have been shown to impact sleep habits. Further, the extent to which there is an effect of gender on the outcome variables or their interactions will be determined.

The expected outcome of this aim is estimates of the effect sizes needed to conduct power analyses for a full-scale study of the associations among glucose excursions, sleep characteristics, and cognitive function, coping, adherence, and adjustment.

Aim 4. Conduct qualitative study using narrative inquiry with all adolescents in our population to identify perceived factors associated with insufficient sleep in adolescents with type 1 diabetes.

In the past several decades, adolescents have shifted to later sleep times, while wake times have remained the same, resulting in insufficient sleep. Barriers to sleep in adolescents include extracurricular activities, work, academics, and social interaction. More recently, electronic media use and video-game playing have been linked to shorter sleep duration. Predictors of disturbed sleep in adolescents and young adults (college students) include emotional and academic stress. Many of these are modifiable behaviors that could be addressed in future interventions. For adolescents with T1D, sleeping late on the weekends has additional risks of hypoglycemic episodes. What is not known are the barriers and facilitators to sleep specific to this population. Interviews will be conducted with adolescents to learn through their stories what are important factors associated with insufficient sleep in this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for at least 6 months

Exclusion Criteria:

* able to comply with protocol

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 youth with type 1 diabetes, age 10-16 years, diagnosed for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Glycemic control | baseline
  Hemoglobin A1C

SECONDARY OUTCOMES:
Executive functioning | baseline
  Trail Making Test Part B

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Grey, DrPH, Principal Investigator — Yale University
Locations (1):
- Yale School of Nursing, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared once analyses are final.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after data collection is complete
Access Criteria: By request to principal investigator